CLINICAL TRIAL: NCT00179023
Title: The Autonomic Nervous System and Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 020548; HL56693
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: OBESITY; HYPERTENSION; PURE AUTONOMIC FAILURE; SHY-DRAGER SYNDROME
Keywords: OBESITY; RESTING ENERGY EXPENDITURE; SYMPATHETIC NERVOUS SYSTEM; HYPERTENSION; AUTONOMIC FAILURE
MeSH Terms: conditions — Obesity; Hypertension; Pure Autonomic Failure; Shy-Drager Syndrome | interventions — Trimethaphan; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 (Other): Estimation of resting energy expenditure and effect of autonomic blockade with trimethaphan infusion.
  Interventions: Drug: Trimethaphan
- Part 2 (closed) (Other): Estimation of autonomic function and effect of autonomic blockade with trimethaphan infusion.
  Interventions: Drug: Trimethaphan
- Part 3 (Other): Estimation of energy metabolism and effect of sympathetic stimulation with pseudoephedrine.
  Interventions: Drug: Pseudoephedrine
- Part 4a (closed) (Other): Isoproterenol sensitivity in adipose and muscle tissue with and without systemic autonomic blockade with trimethaphan infusion.
  Interventions: Drug: Trimethaphan
- Part 4b (closed) (Other): Metabolic and hemodynamic response to submaximal exercise in adipose and muscle tissue with and without systemic autonomic blockade with trimethaphan infusion.
  Interventions: Drug: Trimethaphan

INTERVENTIONS:
Drug: Trimethaphan — Start dose: 0.05 ml/min (0.5 mg/min), IV infusion. The dose will be increased every 2-4 minutes to 1, 2, 4, and 5 mg/min. Total duration: 1 hour
  Arms: Part 1; Part 4a (closed); Part 4b (closed)
Drug: Trimethaphan — Start dose: 0.05 ml/min (0.5 mg/min), IV infusion. The dose will be increased every 30 minutes to 1, 2, 4, and 5 mg/min. Total duration: 1-2 hours
  Arms: Part 2 (closed)
Drug: Pseudoephedrine — 30mg tablet,VO. Single dose.
  Other Names: Sudafed
  Arms: Part 3

SUMMARY:
In its simplest terms, obesity is the results of a positive balance between food intake and energy expenditure (EE). I.e., we take in more energy, in the form of food, than we expend, e.g., by exercise. In our sedentary society, resting EE accounts for most of total energy expenditure. The sympathetic nervous system (SNS, the one that produces adrenaline) is thought to contribute to resting EE. This conclusion is based on experiments where resting EE is decreased by beta-blockers, high blood pressure medicines that block only one aspect of the sympathetic nervous system. The investigators propose to use a different approach, by using a medication called trimethaphan that produces transient withdrawal of the autonomic nervous system. The investigators will then compare the measured resting EE before and after SNS withdraw and quantify the degree of contribution to the resting EE by the SNS and delineate differences between healthy normal, healthy obese, and patients with autonomic dysfunctions.

DETAILED DESCRIPTION:
The rationale for this study is that even small alterations to energy metabolism can significantly change energy balance and body weight in the long term. We will test the hypothesis that the sympathetic nervous system (SNS) activity contributes to resting and thermogenic components of energy expenditure (EE).

This study is divided in four different parts: (1), (2), (3), (4).

Part (1): we will gauge the contribution of the sympathetic nervous system to resting energy expenditure, blood pressure, and determine differences between lean, obese, and patients with primary autonomic failure .

Part (2): we will determine the degree of sympathetic blockade by a gradual infusion of the ganglionic blocker trimethaphan.[Part 2 has been closed]

Part (3): we will determine the energy balance in patients with primary autonomic failure.

Part (4): we will determine the contribution of the sympathetic nervous system to lipolysis.[Part 4 has been closed]

Subjects selections*:

For part (1) and (2) we will study six groups of subjects (n = 40 for each group): patients with pure autonomic failure, patients with multiple system atrophy, healthy normal controls (BMI <= 25), obese controls (BMI 30-40) and obese hypertensive (BMI 30-40) and lean hypertensive (BMI 20-28). A time interval of at least 1 week is required for those subjects who wish to participate in part (1) and part (2). For part (3) we will study two groups of subjects (n=12 for each group): patients with autonomic failure, and their age sex-matched sedentary, healthy controls. For part (4) we will study two groups of subjects (n=12 for each group): healthy normal controls (BMI 20-25), obese controls (BMI 30-40).

*Part 2 and 4 have been closed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal (BMI <= 25 Kg/m2), obese (BMI between 30 and 40)volunteers, lean hypertensive (BMI 20-28 Kg/m2), and obese hypertensive (BMI between 30 and 40)
* Ages 18-60
* Patients with pure autonomic failure and multiple system atrophy ages 18-80, referred to our service for the diagnosis and treatment of their condition, and their age sex-matched sedentary, healthy controls ages 18-80

Exclusion criteria:

* All medical students
* Pregnant women
* Heart failure, symptomatic coronary artery disease, liver impairment, history of stroke or myocardial infarction, glaucoma
* History of serious allergies or asthma
* Subjects using beta-blockers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2003-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in supine systolic blood pressure after achieving complete ganglionic blockade. | 1-2 hour

SECONDARY OUTCOMES:
Change in resting energy expenditure after achieving complete autonomic blockade. | 1-2 hour

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shibao C, Gamboa A, Diedrich A, Ertl AC, Chen KY, Byrne DW, Farley G, Paranjape SY, Davis SN, Biaggioni I. Autonomic contribution to blood pressure and metabolism in obesity. Hypertension. 2007 Jan;49(1):27-33. doi: 10.1161/01.HYP.0000251679.87348.05. Epub 2006 Nov 20. PMID 17116758
- [Result] Shibao C, Buchowski MS, Chen KY, Yu C, Biaggioni I. Chronic sympathetic attenuation and energy metabolism in autonomic failure. Hypertension. 2012 May;59(5):985-90. doi: 10.1161/HYPERTENSIONAHA.111.190157. Epub 2012 Apr 2. PMID 22469621